CLINICAL TRIAL: NCT00741767
Title: The Impact of Salmeterol-Fluticasone on Sleep in Patients With COPD (Advair and Quality of Sleep in COPD)
Brief Title: The Impact of Salmeterol-Fluticasone on Sleep in Patients With COPD
Acronym: AQuOS-COPD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study subject enrollment difficulties
Sponsor: Northwestern University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Ravi Kalhan, Assistant Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 3582
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Obstructive Pulmonary Disease; Sleep Disorders
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Sleep; Sleep quality; Lung hyperinflation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Salmeterol-fluticasone (Other): Patients randomized to receive salmeterol-fluticasone 250/50 twice daily for 4 weeks. Patients will cross-over and receive placebo medication for 4 weeks later in the study.
  Interventions: Drug: salmeterol-fluticasone
- Placebo (Other): Patients randomized to receive placebo medication twice daily for 4 weeks. Patients will cross-over and receive study medication later in the study.
  Interventions: Drug: salmeterol-fluticasone

INTERVENTIONS:
Drug: salmeterol-fluticasone — 250ug salmeterol/50ug fluticasone inhaled via an oral inhaler twice daily
  Other Names: Advair Diskus

SUMMARY:
The purpose of this study is to determine if Advair Diskus improves sleep quality by reducing lung hyperinflation in COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a common and clinically important disease characterized by chronic, irreversible airflow obstruction. Poor sleep quality and insomnia are well described phenomena in patients with COPD. Several studies suggest sleep disturbance adversely affects quality of life and may worsen daytime pulmonary function in COPD patients. Improving sleep quality in patients with COPD, therefore, may not only improve health quality, but also attenuate the decline in daytime pulmonary function.

Previous studies investigating the effects of inhaled bronchodilators on sleep quality in COPD have shown conflicting results. These conflicting data prompted us to perform a retrospective study on patients with COPD and co-existing sleep apnea (OSA) investigating the effects of mechanical lung function impairment and lung hyperinflation on sleep. Our study found a significant correlation between increased lung hyperinflation and reduced sleep efficiency (a measure of sleep quality), and this relationship was preserved in a multivariable regression model.

We hypothesize that Advair Diskus improves sleep quality by reducing lung hyperinflation in COPD. To test this hypothesis, we propose a double-blinded, placebo controlled cross-over study of Advair Diskus in patients with COPD and lung hyperinflation.

It was mutually decided by the sponsor and principal investigator to terminate the study early due to study subject enrollment difficulties.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years of age
* BMI<30
* Former smokers with ≥ 10 pack-year history
* Diagnosis of COPD, as defined by the American Thoracic Society (FEV1/FVC < 70 with history of exposure to noxious particles or gases)
* Moderate to severe COPD as defined as an FEV1 ≤ 80% predicted
* Functional residual capacity > 120% or inspiratory capacity < 80% predicted on pulmonary function testing
* Poor subjective sleep quality: All subjects included must answer "yes" to at least one of the following questions:

  1. Do you have trouble falling asleep?
  2. Do you have trouble staying asleep?
  3. Do you not get enough sleep?
  4. Do you wake up too early and not be able to get back to sleep?
  5. Do you fall asleep during the day?

Exclusion Criteria:

* Conditions that in the judgment of the investigator would interfere with subject participation in the study
* BMI > 30
* History of or physician diagnosed pulmonary disorder other than COPD
* History of significant obstructive sleep disordered breathing (apnea-hypopnea index > 15) or presence of central sleep apnea
* History of narcolepsy, primary hypersomnia, periodic limb movement disorder, or parasomnia
* History of psychiatric illness
* Presence of decompensated heart failure
* Use of prednisone, antibiotic therapy, or new medication for COPD in the previous 3 months
* Use of any sleep aids
* History of ≥ 1 COPD exacerbation (defined as requiring oral corticosteroids and/or antibiotics as either an outpatient or inpatient)
* Known allergy or significant adverse reactions to inhaled beta2-agonists and inhaled corticosteroids (not including thrush and dysphonia)
* Pregnancy or lactating
* Inability or unwillingness to provide informed consent
* Inability to effectively use study medication or perform baseline measurements
* Inability to be contacted by phone

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2010-09 (Estimated); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Changes in subjective measures of sleep quality | 16 weeks
Changes in objective measures of sleep and daytime cognitive function | 16 weeks

SECONDARY OUTCOMES:
Changes in lung hyperinflation and systemic inflammation | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Kalhan, MD, MS, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States